CLINICAL TRIAL: NCT07048275
Title: Exploring the Application of Virtual Reality in Enhancing Chest Percussion Techniques, Reducing Caregiver Stress, and Improving Teaching Effectiveness for Caregivers of Children With Pneumonia
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Head Nurse, National Taiwan University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 202411017RINC
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Virtual Reality

STUDY DESIGN:
Intervention Model Description: The assessment time points are set on the day of hospital admission or transfer (T1), and the fourth day after the teaching intervention (T2). Both the control group and the experimental group will be evaluated using the following questionnaires: Chest Percussion Skill Assessment, Chest Percussion Knowledge Test, Caregiver Stress Self-Assessment Scale, and Pediatric Respiratory Sounds. The experimental group will additionally undergo an evaluation of teaching effectiveness.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Chest Percussion Teaching Program (Experimental): Participants will be assessed at two time points: on the day of hospital admission or transfer, and on the fourth day after the teaching intervention.
  Interventions: Behavioral: Virtual Reality Chest Percussion Teaching Program
- Nurse-Led Chest Percussion Health Education Program (No Intervention): Participants will be assessed at two time points: on the day of hospital admission or transfer, and on the fourth day after the teaching intervention.

INTERVENTIONS:
Behavioral: Virtual Reality Chest Percussion Teaching Program — Participants will be assessed at two time points: on the day of hospital admission or transfer, and on the fourth day after the teaching intervention.
  Arms: Virtual Reality Chest Percussion Teaching Program

SUMMARY:
This study intends to adopt a Randomized Controlled Trial (RCT) design to explore the application of virtual reality in training chest percussion techniques for children with pneumonia. The aim is to evaluate the accuracy and efficiency of caregivers in performing this technique. The study will analyze the potential clinical benefits of improving caregivers' chest percussion skills and reducing caregiver stress

DETAILED DESCRIPTION:
This study explores the application of virtual reality (VR) in training chest percussion techniques for children with pneumonia, aiming to enhance the accuracy and efficiency of caregivers performing this technique. Chest percussion is a critical component of pulmonary physiotherapy, especially for pediatric patients with respiratory diseases requiring adjunctive chest therapy.

The purpose of this paper is to investigate the use of VR technology in chest percussion training, including its underlying principles, clinical practice, and future development. By reviewing both domestic and international research, the study analyzes the potential clinical benefits of improving caregivers' chest percussion skills and alleviating caregiver stress.

Research Objective:

To explore the application of virtual reality in enhancing chest percussion techniques, reducing caregiver stress, and improving teaching effectiveness for caregivers of children with pneumonia.

ELIGIBILITY:
Inclusion Criteria:

- Primary caregivers of pediatric patients who have been diagnosed by a physician as requiring chest percussion as an adjunct therapy and are at least 18 years old

Exclusion Criteria:

1. Severe communication barriers (inability to communicate in Mandarin or Taiwanese, blindness, or deafness) that prevent understanding of the simulator.
2. Primary caregivers of pediatric patients with contraindications to chest percussion therapy, such as rib fractures, osteoporosis, tumors or skin graft sites, or pulmonary embolism.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Pediatric Chest Physiotherapy Technique Assessment Form | Participants will be assessed at two time points: on the day of hospital admission or transfer, and on the fourth day after the teaching intervention
  An evaluation checklist consisting of nine items was developed in accordance with the nursing skills standards for pediatric chest physiotherapy
Pediatric Chest Percussion Knowledge Assessment | Participants will be assessed at two time points: on the day of hospital admission or transfer, and on the fourth day after the teaching intervention
  includes ten items addressing percussion techniques and precautions, and evaluates caregivers' knowledge of the chest percussion process and safety considerations.

SECONDARY OUTCOMES:
Caregiver Stress Self-Assessment Scale | Participants will be assessed at two time points: on the day of hospital admission or transfer, and on the fourth day after the teaching intervention
  The scale consists of 14 items covering aspects such as physical and emotional impact, interpersonal relationships, and financial burden. A 4-point Likert scale is used, with each item scored from 0 to 3. The scoring criteria are as follows: "never" = 0 points, "rarely" = 1 point, "sometimes" = 2 points, and "often" = 3 points. Total scores range from 0 to 42, with scores of 0-13 indicating good adjustment, 14-25 indicating mild caregiver stress, and 26-42 indicating a high level of perceived caregiver stress.
Respiratory Sounds of Pediatric Patients | Participants will be assessed at two time points: on the day of hospital admission or transfer, and on the fourth day after the teaching intervention
  A physician confirmed the presence of abnormal breath sounds in the pediatric patient through auscultation, including crackles (moist rales), rhonchi (dry rales), wheezing, and stridor.
Learning Outcomes of Virtual Reality-Based Teaching Materials | Fourth day after virtual reality intervention
  The instrument includes 10 items, each rated on a 6-point Likert scale, with scores ranging from 0 (strongly disagree) to 5 (strongly agree).

CONTACTS AND LOCATIONS:
Locations (1):
- Hui-Mei, Chen, Yuanlin, Taiwan

IPD SHARING:
Plan to Share IPD: No
Patient privacy consideration